CLINICAL TRIAL: NCT02594085
Title: An Exploratory Study Investigating Adhesive Reaction to Output
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CP261
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Ileostomy
MeSH Terms: interventions — Sugp2 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Patch 3/Patch4 + Patch1/patch2 + patch 5/patch 6 (Experimental): The subjects test 6 adhesive strips; two in each test period. The patches are tested in pairs i.e Patch 1 and patch 2 are a pair; Patch 3 and Patch 4 are a piar and patch 5 and patch 6 are a pair. The test order of the patch pairs is randomised between the three periods.
  In this arm the the subjects test:
  Test period 1: Patch 3 and Patch 4 Test period 2: Patch 1 and Patch 2 Test period 3: Patch 5 and Patch 6
  Interventions: Other: Patch 1; Other: Patch 2; Other: Patch 3; Other: Patch 4; Other: patch 5; Other: Patch 6
- Patch 1/Patch2 + Patch3/patch4 + patch 5/patch 6 (Experimental): The subjects test 6 adhesive strips; two in each test period. The patches are tested in pairs i.e Patch 1 and patch 2 are a pair; Patch 3 and Patch 4 are a piar and patch 5 and patch 6 are a pair. The test order of the patch pairs is randomised between the three periods.
  In this arm the the subjects test:
  Test period 1: Patch 1 and Patch 2 Test period 2: Patch 3 and Patch 4 Test period 3: Patch 5 and Patch 6
  Interventions: Other: Patch 1; Other: Patch 2; Other: Patch 3; Other: Patch 4; Other: patch 5; Other: Patch 6
- Patch 1/Patch2 + Patch5/patch 6 + patch 3/patch 4 (Experimental): The subjects test 6 adhesive strips; two in each test period. The patches are tested in pairs i.e Patch 1 and patch 2 are a pair; Patch 3 and Patch 4 are a piar and patch 5 and patch 6 are a pair. The test order of the patch pairs is randomised between the three periods.
  In this arm the the subjects test:
  Test period 1: Patch 1 and Patch 2 Test period 2: Patch 3 and Patch 4 Test period 3: Patch 5 and Patch 6
  Interventions: Other: Patch 1; Other: Patch 2; Other: Patch 3; Other: Patch 4; Other: patch 5; Other: Patch 6
- Patch 3/Patch4 + Patch5/patch6 + patch 3/patch 4 (Experimental): The subjects test 6 adhesive strips; two in each test period. The patches are tested in pairs i.e Patch 1 and patch 2 are a pair; Patch 3 and Patch 4 are a piar and patch 5 and patch 6 are a pair. The test order of the patch pairs is randomised between the three periods.
  In this arm the the subjects test:
  Test period 1: Patch 3 and Patch 4 Test period 2: Patch 5 and Patch 6 Test period 3: Patch 1 and Patch 2
  Interventions: Other: Patch 1; Other: Patch 2; Other: Patch 3; Other: Patch 4; Other: patch 5; Other: Patch 6
- Patch 5/Patch 6 + Patch 3/patch 4 + patch 1/patch 2 (Experimental): The subjects test 6 adhesive strips; two in each test period. The patches are tested in pairs i.e Patch 1 and patch 2 are a pair; Patch 3 and Patch 4 are a piar and patch 5 and patch 6 are a pair. The test order of the patch pairs is randomised between the three periods.
  In this arm the the subjects test:
  Test period 1: Patch 5 and Patch 6 Test period 2: Patch 3 and Patch 4 Test period 3: Patch 1 and Patch 2
  Interventions: Other: Patch 1; Other: Patch 2; Other: Patch 3; Other: Patch 4; Other: patch 5; Other: Patch 6
- Patch 5/Patch 6 + Patch1/patch2 + patch 3/patch 4 (Experimental): The subjects test 6 adhesive strips; two in each test period. The patches are tested in pairs i.e Patch 1 and patch 2 are a pair; Patch 3 and Patch 4 are a piar and patch 5 and patch 6 are a pair. The test order of the patch pairs is randomised between the three periods.
  In this arm the the subjects test:
  Test period 1: Patch 1 and Patch 2 Test period 2: Patch 3 and Patch 4 Test period 3: Patch 5 and Patch 6
  Interventions: Other: Patch 1; Other: Patch 2; Other: Patch 3; Other: Patch 4; Other: patch 5; Other: Patch 6

INTERVENTIONS:
Other: Patch 1 — Patch 1 describes a test system which contains an adhesive strip and an adhesive patch with a sleeve. The sleeve of Patch 1 contains the subjects own feces. The Patch is placed over the adhesive strip to investigate the impact of output on the adhesive strip
Other: Patch 2 — Patch 2 describes a test system which contains an adhesive strip and an adhesive patch with a sleeve. The sleeve Patch 2 contains the subjects own feces and filler. The Patch is placed over the adhesive strip to investigate the impact of output on the adhesive strip
Other: Patch 3 — Patch 3 describes a test system which contains an adhesive strip and an adhesive patch with a sleeve. The sleeve of Patch 3 contains simulated output. The Patch is placed over the adhesive strip to invesitgate the impact of output on the adhesive strip
Other: Patch 4 — Patch 4 describes a test system which contains an adhesive strip and an adhesive patch with a sleeve. The sleeve of Patch 4 contains simulated output with filler. The Patch is placed over the adhesive strip to investigate the impact of output on the adhesive strip
Other: patch 5 — Patch 5 describes a test system which contains an adhesive strip and an adhesive patch with a sleeve. The sleeve of Patch 5 contains buffer. The Patch is placed over the adhesive strip to investigate the impact of output on the adhesive strip
Other: Patch 6 — Patch 6 describes a test system which contains an adhesive strip and an adhesive patch with a sleeve. The sleeve of Patch 6 contains buffer with filler. The Patch is placed over the adhesive strip to investigate the impact of output on the adhesive strip

SUMMARY:
The objective is to investigate the impact that faecal output has on adhesives.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had an ileostomy for more than 3 months
4. Have intact skin on the area used in the evaluation
5. Has an ileostomy with a diameter (≤) 35mm

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal area
5. Convex user
6. Participate in other interventional clinical investigations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Remaining adherent area of the adhesive | 8 hours
  The remaining adherent area of the adhesive strips is assessed by measuring the difference in total area of output and swelling.

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Medical Director
Locations (1):
- Coloplast A/S, Humlebæk, Denmark